CLINICAL TRIAL: NCT00983957
Title: The Effect of the Co-administration of BMS-790052 on the Pharmacokinetics of a Combined Oral Contraceptive Containing Ethinyl Estradiol and Norgestimate (Ortho Tri-Cyclen®) in Healthy Female Subjects
Brief Title: Study to Assess the Effect of BMS-790052 on the Pharmacokinetics of Ortho Tri-Cyclen® in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AI444-020
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2015-09-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — daclatasvir; norgestimate, ethinyl estradiol drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-790052 plus Ortho Tri-Cyclen® (Experimental)
  Interventions: Drug: BMS-790052; Drug: Ortho Tri-Cyclen®

INTERVENTIONS:
Drug: BMS-790052 — Tablets, Oral, 60 mg, once daily, 10 days
Drug: Ortho Tri-Cyclen® — Tablets, Oral, once daily, 78 days

SUMMARY:
The purpose of this study is to assess the effect of BMS-790052 on the pharmacokinetics of Ortho Tri-Cyclen® in healthy female subjects.

ELIGIBILITY:
Key Inclusion Criteria:

* Healthy female subjects, 18-45 years, BMI 18-32 kg/m².
* Must be using an adequate method of contraception to avoid pregnancy throughout the study.

Key Exclusion Criteria:

* Abnormal Pap smear within 1 yr of dosing, and abnormal menstrual cycle during the 3 months prior to enrollment.
* Any significant or chronic uncontrolled medical illness.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2009-10; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- United States (2):
  - MDS Pharma Services (US), Inc, Tempe, Arizona
  - Covance Clinical Research Unit, Inc., Austin, Texas
- Local Institution, Saint-Laurent, Quebec, Canada

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 47 participants were enrolled; 20 were treated. Reasons 27 participants were not treated: 21 no longer met study criteria, 2 withdrew consent, and 4 other reasons.
Groups:
- Ortho Tri-Cyclen + Daclatasvir: Participants received sequentially Treatment A: Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily up to Day 28, Treatment B: Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 29 to 56 and Treatment C: Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 57 to 77 concomitantly with daclatasvir, two tablets of 30-mg, orally, once daily from Day 68 to 77.
Period: Overall Study
Arm/Group | Ortho Tri-Cyclen + Daclatasvir
Started | 20
Treatment A | 20
Treatment B | 20
Treatment C | 18
Completed | 18
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Personal Reasons | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Arm/Group | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.8 (7.36)
Age, Customized [Number; unit: participants]
  <= 45 years | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Ethinyl Estradiol
Description: Ethinyl Estradiol is an analyte of Ortho Tri-Cyclen. Ethinyl Estradiol was measured in plasma, using liquid chromatography-tandem mass spectrometry (LC-MS/MS) by a validated analytical method during the period of known analyte stability. Cmax was measured in picograms per milliliter (pg/mL) and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 hours post-dose on Days 49 and 77
Population: All participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picogram per millilitre (pg/mL)
Groups:
- Ortho Tri-Cyclen: Treatment B: Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 29 to 56.
- Ortho Tri-Cyclen + Daclatasvir: Treatment C: Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 57 to 77 concomitantly with daclatasvir, two tablets of 30-mg, orally, once daily from Day 68 to 77.
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
picogram per millilitre (pg/mL) | 118.53 (34) | 134.70 (30)
Statistical Analysis 1: Comparison: Ortho Tri-Cyclen vs Ortho Tri-Cyclen + Daclatasvir; Mixed effect models were fitted to log-transformed data with treatment as a fixed effect, and measurements within each participant as repeated measurements; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.105, 90% CI 2-sided [1.023 to 1.195] — Point estimates and 90% Confidence Interval (CIs) for treatment differences on the log scale were exponentiated to obtain estimates for ratios of geometric means on the original scale

2. Secondary Outcome: Maximum Observed Plasma Concentration of Norgestrel
Description: Norgestrel is an NGM metabolite and was measured in plasma using liquid chromatography-mass spectrometry by a validated analytical method during the period of known analyte stability. Cmax was measured in picograms per milliliter (pg/mL) and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose on Days 49 and 77
Population: All participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
pg/mL | 2674.69 (32) | 2815.98 (32)
Statistical Analysis 1: Comparison: Ortho Tri-Cyclen vs Ortho Tri-Cyclen + Daclatasvir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.071, 90% CI 2-sided [0.988 to 1.160] — Point estimates and 90% CIs for treatment differences on the log scale were exponentiated to obtain estimates for ratios of geometric means on the original scale

3. Primary Outcome: Area Under the Concentration-Time Curve (AUC) in 1 Dosing Interval of Ethinyl Estradiol
Description: Ethinyl Estradiol was measured in plasma, using liquid chromatography-tandem mass spectrometry by a validated analytical method during the period of known analyte stability. AUC(TAU) was measured in picograms multiplied by hours (h) per milliliter (pg*h/mL) and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose on Days 49 and 77
Population: All participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
pg*h/mL | 959.37 (38) | 994.40 (35)
Statistical Analysis 1: Comparison: Ortho Tri-Cyclen vs Ortho Tri-Cyclen + Daclatasvir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted geometric mean = 1.009, 90% CI 2-sided [0.951 to 1.070] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Area Under the Concentration-Time Curve in 1 Dosing Interval of Norgestrel
Description: Norgestrel was measured in plasma, using liquid chromatography-tandem mass spectrometry by a validated analytical method during the period of known analyte stability. AUC(TAU) was measured in picograms multiplied by hours (h) per milliliter (pg*h/mL) and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose on Days 49 and 77
Population: All participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*h/mL
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
pg*h/mL | 47258.35 (38) | 51760.43 (35)
Statistical Analysis 1: Comparison: Ortho Tri-Cyclen vs Ortho Tri-Cyclen + Daclatasvir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.121, 90% CI 2-sided [1.018 to 1.234] — [estimate comment as in outcome 2, analysis 1]

5. Secondary Outcome: Time of Maximum Observed Plasma Concentration of Norgestrel
Description: Norgestrel was measured in plasma, using liquid chromatography-tandem mass spectrometry by a validated analytical method during the period of known analyte stability. Tmax was measured in hours (h), and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose on Days 49 and 77
Population: All participants who received the study drug.
Measure: Median (Full Range); unit: hours
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
hours | 1.8 [1.0 to 3.0] | 2.0 [1.0 to 8.0]

6. Primary Outcome: Time of Maximum Observed Plasma Concentration of Ethinyl Estradiol
Description: Ethinyl Estradiol was measured in plasma, using liquid chromatography-tandem mass spectrometry by a validated analytical method during the period of known analyte stability. Tmax was measured in hours (h), and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose on Days 49 and 77
Population: All participants who received the study drug
Measure: Median (Full Range); unit: hours
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
hours | 1.5 [1.0 to 2.0] | 1.5 [1.0 to 2.0]

7. Primary Outcome: Maximum Observed Plasma Concentration of Norelgestromin
Description: Norelgestromin is a major active metabolite of norgestimate (NGM) which is found in Ortho Tri-Cyclen. Norelgestromin was measured in plasma, using liquid chromatography-tandem mass spectrometry by a validated analytical method during the period of known analyte stability. Cmax was measured in nanograms per milliliter (ng/mL) and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose on Days 49 and 77
Population: All participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per millilitre (ng/mL)
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
nanogram per millilitre (ng/mL) | 1.99 (20) | 2.10 (20)
Statistical Analysis 1: Comparison: Ortho Tri-Cyclen vs Ortho Tri-Cyclen + Daclatasvir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.059, 90% CI 2-sided [0.988 to 1.135] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, and Who Died
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not have a causal relationship with treatment. SAE=a medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Time Frame: For AEs from start of treatment (Day 1) up to Day 78 or discharge and for SAEs from Day 1 to 30 days after last dose of study drug
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
participants
  SAE | 0 | 0
  AE Leading to Discontinuation | 0 | 1
  Death | 0 | 0

9. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory marked abnormalities were defined as Hematocrit (low) as <0.85*Pre-treatment (PreRx), Hemoglobin (low) as <0.85*PreRx, Aspartate Aminotransferase (AST) (high) as >1.25*PreRx if PreRx > upper limits of normal (ULN); >1.25*ULN if PreRx <=ULN; >1.25*ULN if PreRx = Missing, Blood in urine (high) as ≥2 PreRx if PreRx ≥1; ≥2 if PreRx <1; ≥2 if PreRx = Missing.
Time Frame: From start of treatment (Day 1) up to Day 78 or discharge
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
participants
  Hematocrit | 1 | 0
  Hemoglobin | 1 | 0
  AST | 1 | 0
  Blood in Urine | 0 | 1

10. Secondary Outcome: Number of Participants Demonstrating a Clinically Meaningful Effect in Vital Signs
Description: Vital Signs were measured after the participant was seated quietly for at least 5 minutes and included systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature. Baseline = Last non-missing pretreatment value.
Time Frame: Baseline, Day 28, Day 29, Day 67, Day 68, Day 78, Day of discharge
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
participants | 0 | 0

11. Secondary Outcome: Number of Participants Demonstrating a Clinically Meaningful Effect in ECG Parameters
Description: The electrocardiogram (ECG) evaluations were performed within ± 15 minutes of the relative time points. ECGs were recorded after the participants were in supine position for at least 5 minutes. ECG parameters measured were: PR interval, QRS complex, QT interval and corrected QT (QTc).
Time Frame: Screening, Day 1, Day 67, Day 77
Population: All participants who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
participants | 0 | 0

12. Primary Outcome: Area Under the Concentration-Time Curve in 1 Dosing Interval of Norelgestromin
Description: Norelgestromin was measured in plasma, using liquid chromatography-tandem mass spectrometry by a validated analytical method during the period of known analyte stability. AUC(TAU) was measured in nanograms multiplied by hours (h) per milliliter (ng*h/mL) and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose on Days 49 and 77
Population: All participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
ng*h/mL | 15.38 (24) | 16.84 (20)
Statistical Analysis 1: Comparison: Ortho Tri-Cyclen vs Ortho Tri-Cyclen + Daclatasvir; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Adjusted geometric mean ratio = 1.115, 90% CI 2-sided [1.063 to 1.171] — [estimate comment as in outcome 2, analysis 1]

13. Primary Outcome: Time of Maximum Observed Plasma Concentration of Norelgestromin
Description: Norelgestromin was measured in plasma, using liquid chromatography-tandem mass spectrometry by a validated analytical method during the period of known analyte stability. Tmax was measured in hours (h), and derived from 24 hour plasma concentration versus time data using non-compartmental methods. Pre-dose concentrations and concentrations prior to the first quantifiable concentration that were below the lower limit of quantitation were treated as missing.
Time Frame: Pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24 h post-dose on Days 49 and 77
Population: All participants who received the study drug.
Measure: Median (Full Range); unit: hours
Arm/Group | Ortho Tri-Cyclen | Ortho Tri-Cyclen + Daclatasvir
Number analyzed (Participants) | 20 | 18
hours | 1.3 [1.0 to 3.0] | 1.5 [1.0 to 2.0]

ADVERSE EVENTS:
Time Frame: From start of treatment (Day 1) up to Day 78 or discharge
Description: On-Treatment Period
Groups:
- All Treated Participants: Participants received sequentially Treatment A: Ortho Tri-Cyclen (OTC) fixed dose combination tablet, orally, once daily up to Day 28, Treatment B: Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 29 to 56 and Treatment C: Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 57 to 77 along with daclatasvir, two tablets of 30-mg, orally, once daily from Day 68 to 77.
- Ortho Tri-Cyclen Days 1-28: Participants received Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily up to Day 28.
- Ortho Tri-Cyclen Days 29-46: Participants received Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 29 to 46.
- Ortho Tri-Cyclen Days 47-56: Participants received Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 47 to 56.
- Ortho Tri-Cyclen Days 57-67: Participants received Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 57 to 67.
- Ortho Tri-Cyclen + Daclatasvir Days 68-77: Participants received Ortho Tri-Cyclen fixed dose combination tablet, orally, once daily from Day 57 to 67 along with daclatasvir two tablets of 30-mg, orally, once daily from Day 68 to 77.
Arm/Group | All Treated Participants | Ortho Tri-Cyclen Days 1-28 | Ortho Tri-Cyclen Days 29-46 | Ortho Tri-Cyclen Days 47-56 | Ortho Tri-Cyclen Days 57-67 | Ortho Tri-Cyclen + Daclatasvir Days 68-77
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 16/20 | 8/20 | 3/20 | 7/20 | 5/18 | 12/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Treated Participants (N=20) | Ortho Tri-Cyclen Days 1-28 (N=20) | Ortho Tri-Cyclen Days 29-46 (N=20) | Ortho Tri-Cyclen Days 47-56 (N=20) | Ortho Tri-Cyclen Days 57-67 (N=18) | Ortho Tri-Cyclen + Daclatasvir Days 68-77 (N=18)
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 0 | 0 | 3
Breast pain (Reproductive system and breast disorders) | 1 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 6 | 5 | 1 | 1 | 0 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vessel puncture site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1 | 0 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 3 | 0 | 0 | 2 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0 | 4
Eye pain (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 9 | 4 | 2 | 6 | 0 | 3
Menstruation irregular (Reproductive system and breast disorders) | 3 | 2 | 0 | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 1 | 0 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 1
Back injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.